CLINICAL TRIAL: NCT02865876
Title: Effectiveness of Corneal Accelerated Crosslinking Versus Conventional Treatment for Infectious Keratitis
Brief Title: Effectiveness of Corneal Accelerated Crosslinking for Infectious Keratitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Collaborators: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI-2015/01/02
Record Dates: First submitted 2016-08-01; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Keratitis
Keywords: Infectious keratitis; Cross-linking
MeSH Terms: conditions — Keratitis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Accelerated Corneal Cross-linking (Experimental): Cross-linking in the management of microbial keratitis is an adjunctive therapy.This procedure is conducted under sterile conditions in the operating room. Tetracaine hydrochloride 0.5% (Ponti Ofteno, Sophia, Mexico) eye drops is apply for topical anesthesia. The corneal epithelium on the edge of the ulcer is cautiously removed using a microsponge. As photosensitizer, riboflavin 0.1% (Vibex, Avedro Inc, Waltham, USA) is used for 10 minutes. After impregnation, the participant´s cornea is irradiaded with UVA-light (370 nm) using 30 mW/cm2 for 3 minutes (which corresponds to a total dose of 5.4J/cm2) with accelerated cross-linking (Avedro Inc., Waltham, USA). After procedure, conventional treatment for keratitis remains unchanged.
  Interventions: Procedure: Accelerated Corneal Cross-linking
- Sham Accelerated Corneal Cross-linking (Sham Comparator): Placebo surgery. This procedure is conducted under sterile conditions in the operating room. Tetracaine hydrochloride 0.5% (Ponti Ofteno, Sophia, Mexico) eye drops is apply for topical anesthesia. Investigators do not perform removal of the corneal epithelium in edge of the ulcer. The researchers conducted "the impregnation phase" applying drops of saline solution for 10 minutes. After impregnation fase, a device is placed in Avedro equipment off (Avedro Inc, Waltham, USA) this device emits white light for 3 minutes. After procedure, conventional treatment for keratitis remains unchanged.
  Interventions: Procedure: Accelerated Corneal Cross-linking

INTERVENTIONS:
Procedure: Accelerated Corneal Cross-linking — All participants in this group receiving conventional therapy (moxifloxacin 0,5% for bacterial keratitis or natamycin for mycotic keratitis) plus accelerated cross-linking (Avedro Inc., Waltham, USA) under topical anesthesia using 0.1% riboflavin (Vibex, Avedro Inc, Waltham, USA) for 10 minutes and irradiation 30 mW/cm2 during 3 minutes.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of accelerated cross-linking (Avedro Inc., Waltham, USA) in the management of microbial keratitis as adjunctive therapy.

DETAILED DESCRIPTION:
Investigators perform a comprehensive ophthalmological examination, including evaluation of risk factors (immunosuppressive status, ocular trauma, previous ocular surgery, contact lens wear, topical corticosteroids use), best-corrected visual acuity (Snellen chart), slit-lamp biomicroscopy, tonometry and fundoscopy. In addition, anterior segment optical coherence tomography imaging (Visante, Carl Zeiss Meditec, Dublin, California, USA), corneal scrapes, culture and clinical photographs at day 1, day 7, month 1 and 3 will be analyzed.

Each participant will be assigned to one of four groups after randomization. Group 1: Initial ulcer on treatment with antibiotic plus sham (n = 66), these partcipants will receive only topical moxifloxacin 0,5% (Vigamoxi, Alcon, Texas, USA) and sham CXL; Group 2: Initial ulcer on treatment with antibiotic plus cross-linking (CXL) (n = 66) receive moxifloxacin plus CXL (riboflavin 0.1% during 10 minutes and irradiation 30 mW/cm2 during 3 minutes using accelerated CXL); Group 3: Refractory corneal ulcer on treatment with antibiotic plus sham (n=66), receive only topical antibiotic plus sham CXL; Group 4: Refractory corneal ulcer on treatment with antibiotic plus CXL will receive their standard medications plus CXL.

Statistical analysis will be divided into four phases: 1) Analysis of compliance, 2) Intention to treat, 3) Losses to follow-up and 4) Variable-response (healing) using Stata/MP 12.0 (Stata Corp., College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with infectious keratitis (initial or refractory to treatment) including bacterial or mycotic keratitis with size larger than 3 mm

Exclusion Criteria:

* herpetic keratitis
* Acanthamoeba keratitis
* pregnancy
* endophthalmitis
* systemic immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Healing | Three months
  Full epithelialization without evidence of infiltrates

SECONDARY OUTCOMES:
Complications | Three months
  Complications associated with accelerated corneal cross-linking, such as corneal perforation or progression

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Graue-Hernandez, MSc, Study Chair — Instituto de Oftalmologia Fundacion Conde de Valenciana
Locations (1):
- Instituto de Oftalmologia Conde de Valenciana, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Investigators describe demographic characteristics of the participants, such as age, gender, etiology, intervention group and the response variables, complications and corneal healing.

REFERENCES:
- [Result] Li Z, Jhanji V, Tao X, Yu H, Chen W, Mu G. Riboflavin/ultravoilet light-mediated crosslinking for fungal keratitis. Br J Ophthalmol. 2013 May;97(5):669-71. doi: 10.1136/bjophthalmol-2012-302518. Epub 2013 Jan 26. No abstract available. PMID 23355529
- [Result] Moren H, Malmsjo M, Mortensen J, Ohrstrom A. Riboflavin and ultraviolet a collagen crosslinking of the cornea for the treatment of keratitis. Cornea. 2010 Jan;29(1):102-4. doi: 10.1097/ICO.0b013e31819c4e43. PMID 19730094
- [Result] Anwar HM, El-Danasoury AM, Hashem AN. Corneal collagen crosslinking in the treatment of infectious keratitis. Clin Ophthalmol. 2011;5:1277-80. doi: 10.2147/OPTH.S24532. Epub 2011 Sep 7. PMID 21966201
- [Result] Price MO, Tenkman LR, Schrier A, Fairchild KM, Trokel SL, Price FW Jr. Photoactivated riboflavin treatment of infectious keratitis using collagen cross-linking technology. J Refract Surg. 2012 Oct;28(10):706-13. doi: 10.3928/1081597X-20120921-06. PMID 23062001
- [Result] Alio JL, Abbouda A, Valle DD, Del Castillo JM, Fernandez JA. Corneal cross linking and infectious keratitis: a systematic review with a meta-analysis of reported cases. J Ophthalmic Inflamm Infect. 2013 May 29;3(1):47. doi: 10.1186/1869-5760-3-47. PMID 23718849
- [Result] Uddaraju M, Mascarenhas J, Das MR, Radhakrishnan N, Keenan JD, Prajna L, Prajna VN. Corneal Cross-linking as an Adjuvant Therapy in the Management of Recalcitrant Deep Stromal Fungal Keratitis: A Randomized Trial. Am J Ophthalmol. 2015 Jul;160(1):131-4.e5. doi: 10.1016/j.ajo.2015.03.024. Epub 2015 Apr 1. PMID 25841317
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558